CLINICAL TRIAL: NCT07110311
Title: Effects of Pet Cats on Nasal and Intestinal Microorganisms in Patients With Allergic Rhinitis Who Are Allergic to Cat Allergen
Brief Title: Impact of Pet Cats on Nasal and Gut Microbiota in Patients With Cat Allergen Allergy
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-797
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — elbow venous blood: 2ml, feces: 5ml, saliva:2ml, tonsil microorganism:2ml, nasal exfoliated cells:2ml, nasal microorganism:2ml.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AR patients with cat ownership.
- AR patients without cat ownership.

SUMMARY:
It has been reported that the incidence of allergic rhinitis (AR) is as high as 24.1% in adults and 16.8% in children in China. A study explored the changes in the incidence of AR in China, and the study showed that the incidence of AR in many cities in China increased significantly from 2005 to 2011. The latest Chinese guidelines for the diagnosis and treatment of allergic rhinitis pointed out that AR is an independent risk factor for asthma, and 40% of AR patients can be complicated with asthma. CARRAD reported that in adult asthma patients who received skin prick test or serum specific IgE (sIgE) for allergens, The positive rates of at least one allergen were 65.4% and 75.4%, respectively. With the acceleration of urbanization and the improvement of people's economic level, more and more families keep pets. Pets can promote people's physical and mental health, but there are also more and more people who are allergic to pets. Some studies have shown that pets are the third major allergen of respiratory allergic diseases, next to dust mites and pollen. Cats are by far one of the most popular pets, but in recent years, the prevalence of cat allergen has gradually increased. Animal allergens are present in saliva, urine, and dander, and they spread into the environment by adhering to the hair and dander of the animals, such that even in homes without pets, the level of allergens in the environment is sufficient to sensitize people. However, at present, the microbial impact of the microorganisms carried by pet cats on their owners and the living environment is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients with moderate to severe dust mite allergic rhinitis were diagnosed based on clinical history and positive cat allergen sensitization tests (skin prick test and/or specific IgE).
* Patients who visited the Department of Otolaryngology of the First Affiliated Hospital of Nanjing Medical University.

Exclusion Criteria:

* Patients who refused to accept specimen and questionnaire collection.
* Patients who had nasal diseases other than allergic rhinitis, such as nasal papilloma and nasal malignant tumor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cat-allergic rhinitis in the Department of Otolaryngology of the First Affiliated Hospital of Nanjing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Metagenomic Sequencing | 3 years
  Metagenomic sequencing was performed on the collected patient samples, cat fecal samples, and environmental samples to obtain relevant information about the microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, PhD, Study Chair — The First Affiliated Hospital, Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu 210000, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No